CLINICAL TRIAL: NCT01165060
Title: Effect of Bezafibrate on Very Long Chain Fatty Acid Metabolism in Men With X-linked Adrenoleukodystrophy (X-ALD)
Brief Title: The Effect of Bezafibrate on the Level of Very Long Chain Fatty Acids (VLCFA) in X-linked Adrenoleukodystrophy (X-ALD)
Acronym: BEZA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: The Stop ALD Foundation (Unknown)
Responsible Party: Department of (pediatric) neurology, Academisch Medisch Centrum, Amsterdam, The Netherlands
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC 09/278
Record Dates: First submitted 2010-07-13; First posted 2010-07-19 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2010-07

CONDITIONS: X-linked Adrenoleukodystrophy; Adrenomyeloneuropathy
Keywords: X-ALD; AMN; adrenomyeloneuropathy phenotype
MeSH Terms: conditions — Adrenoleukodystrophy | interventions — Bezafibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bezafibrate (Experimental): All patients in the trial will use bezafibrate 400 mg once daily until week 12, and subsequently use 800 mg onde daily until week 24.
  Interventions: Drug: Bezafibrate

INTERVENTIONS:
Drug: Bezafibrate — Week 0 to 12: 400 mg once daily 1 tablet. Week 13 to 24: 400 mg once daily 2 tablets.
  Other Names: Bezalip retard.

SUMMARY:
X-linked adrenoleukodystrophy (X-ALD) is an inherited metabolic disorder characterised by accumulation of very long chain fatty acids (VLCFA) in plasma and tissue. Presumably this accumulation is responsible for tissue damage. The disease can cause severe demyelinisation of the central nervous system usually causing death in childhood or progressive ambulatory problems in adults caused by a progressive myelopathy. For the latter category of patients no curative treatment is currently available. Recent investigations in human fibroblasts and mice identified bezafibrate as an agent that might reduce VLCFA in patients with X-ALD.

Objective of the study:

The trial is designed as an open-label pilot study. The main goal is to investigate if bezafibrate can reduce VLCFA in vivo in patient with X-ALD. If there is indeed a biochemical effect, a large follow-up study will be initiated with clinical outcome parameters.

Study design:

10 men with X-ALD will use bezafibrate during a period of 6 months (in combination with a low fat diet). On 6 different time points the participants will undergo a venipuncture for detecting possible side effects and to determine the biochemical outcome parameters.

Study population:

Adult men with X-linked adrenoleukodystrophy.

Intervention (if applicable):

Bezafibrate.

Primary study parameters/outcome of the study:

The primary outcome parameters are cholesterol levels (total-, LDL, and HDL) and levels of triglycerides in plasma, VLCFA levels in plasma, leukocytes and erythrocytes and also C26:0-lyso-PC in bloodspots.

Secondary study parameters/outcome of the study (if applicable):

Secondary outcome parameters are side-effects (subjective and abnormalities in the safety lab).

ELIGIBILITY:
Inclusion Criteria:

* an age of 18 years or older
* capable of giving informed consent and capable of visiting the hospital for follow-up visits
* no contra-indications for the use of bezafibrate, e.g. kidney- and/or liver disease.
* confirmed X-ALD, AMN phenotype (confirmed by VLCFA analysis or analysis of the ABCD1 gene)

Exclusion Criteria:

* use of medication that lowers cholesterol and/or triglycerides (e.g. statins)
* liver disease or and increase in serum CK of more than 3 times the baseline level
* treatment with Lorenzo's oil in the 8 weeks preceding the trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Very long chain fatty acids (VLCFA; C22:0, C24:0 and C26:0) in plasma, lymphocytes and erythrocytes. | 24 weeks

SECONDARY OUTCOMES:
Side effects | At 4, 8, 12, 16, 20 and 24 weeks.
Cholesterol (total-, HDL, and LDL-cholesterol) in plasma. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bwee Tien Poll - The, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academisch Medisch Centrum, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Engelen M, Tran L, Ofman R, Brennecke J, Moser AB, Dijkstra IM, Wanders RJ, Poll-The BT, Kemp S. Bezafibrate for X-linked adrenoleukodystrophy. PLoS One. 2012;7(7):e41013. doi: 10.1371/journal.pone.0041013. Epub 2012 Jul 20. PMID 22911730